CLINICAL TRIAL: NCT01364766
Title: The Impact of Continuous Glucose Monitor Use in the Classroom/School Environment
Brief Title: Continuous Glucose Monitor Use in School
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tandy Aye, Assistant Professor, Stanford University
Other Study IDs: SU-08122010-6709
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find the impact of continuous blood glucose sensors use in the classroom/school environment. We will be asking the subject,subject's parent and subject's teachers to complete a short survey/questionnaire. The survey will take approximately 10-15 minutes.

DETAILED DESCRIPTION:
The purpose of this study is to find the impact of continuous blood glucose sensors use in the classroom/school environment. Recent technological advancements in diabetes management have resulted in increased use of devices during class/school. Although many studies have examined the quality of life and the impact on the family and subject of these devices, to our knowledge this is the first study that will examine the impact of the continuous glucose monitor during class/school. To our knowledge, this is first study to involve the teachers. The results of this study is particularly important since the future of diabetes therapy will be to use continuous glucose monitors and insulin pumps to develop a closed loop system of insulin therapy or "artificial pancreas."

ELIGIBILITY:
Inclusion Criteria:

Diabetes use continuous glucose monitor in school

Exclusion Criteria not using a continuous glucose monitor

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Anyone with diabetes mellitus who is wearing a continous glucose sensor and is in school.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
CGM usefulness score | 1 yr

SECONDARY OUTCOMES:
Diabetes Comfort score | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benassi K, Drobny J, Aye T. Real-time continuous glucose monitoring systems in the classroom/school environment. Diabetes Technol Ther. 2013 May;15(5):409-12. doi: 10.1089/dia.2012.0314. Epub 2013 Mar 26. PMID 23530577